CLINICAL TRIAL: NCT04969367
Title: Measuring Physical Activity in Transfusion Dependent Patients With Myelodysplastic Syndrome (MDS)
Brief Title: Physical Activity in Transfusion Dependent Patients With Myelodysplastic Syndrome
Status: Withdrawn | Type: Observational
Why Stopped: Staffing
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: 21D.214; JT 16333 (Other: JeffTrial Number)
Record Dates: First submitted 2021-07-06; First posted 2021-07-20 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (activity monitor): Patients wear an activity monitor (Fitbit) for 90 days. Patients also undergo collection of blood samples and complete questionnaires twice weekly for up to 90 days.
  Interventions: Other: Medical Device Usage and Evaluation; Procedure: Biospecimen Collection; Other: Questionnaire Administration; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Medical Device Usage and Evaluation — Wear activity monitor (Fitbit)
Procedure: Biospecimen Collection — Undergo collection of blood samples
Other: Questionnaire Administration — Complete questionnaires
Other: Quality-of-Life Assessment — Complete questionnaires

SUMMARY:
This study assesses feasibility and patient acceptability of using a Fitbit to monitor step count and heart rate in transfusion dependent patients with myelodysplastic syndrome. Information from this study may help researchers understand if there is any correlation between activity level and anemia.

DETAILED DESCRIPTION:
This study assesses feasibility and patient acceptability of using a Fitbit to monitor step count and heart rate in transfusion dependent patients with myelodysplastic syndrome. Information from this study may help researchers understand if there is any correlation between activity level and anemia.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed pathologic diagnosis of MDS
* Requiring >= 2 blood transfusions in the past month if previously diagnosed or hemoglobin =< 8 g/dL if newly diagnosed
* Age >= 18
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Ambulatory (use of a walking aid, such as a cane or rollator, is acceptable)
* Able to give informed consent
* Willing to comply with all study procedures and available for the duration of the study
* Able to read and/or understand English
* Have access to an iPhone 4S or later, iPad 3 generation or later, Android 5.0 or later, or Windows 10 device
* Have access to Bluetooth low energy (LE) and internet connection for syncing

Exclusion Criteria:

• Uncontrolled illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with myelodysplastic syndrome (MDS) recruited from the Department of Medical Oncology- Jefferson Health
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
Accrual rate | Up to 90 days
  accrual rate will be measured by counting subjects
Acceptability | Up to 90 days
  Acceptability will be measured by a short survey
compliance with device | Up to 90 days
  compliance with device (80% of the 90-day intervention time)
retention rate | Up to 90 days
  retention rate of subjects will be measured by counting at 90 days
Acceptability | Up to 90 days
  Acceptability will be measured by an interview addressing participant satisfaction

SECONDARY OUTCOMES:
Daily step count | Up to 90 days
  Daily step count
Average daily resting heart rate | Up to 90 days
  average daily resting heart rate
Fact-An score (assessed twice a week), | Up to 90 days
  Fact-An score (assessed twice a week),
Hemoglobin level measured by CBC twice a week | Up to 90 days
  Hemoglobin level measured by CBC twice a week

CONTACTS AND LOCATIONS:
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/67/NCT04969367/Prot_SAP_001.pdf